CLINICAL TRIAL: NCT01846559
Title: Study of the Effect of Ticagrelor and Clopidogrel on the Immune Response of Healthy Volunteers
Brief Title: The Antiplatelet and Immune Response Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STH17062
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Immune system processes
MeSH Terms: interventions — Endotoxins; Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Clopidogrel & Endotoxin (Experimental): Clopidogrel (tablet) over 8 days Day 1: 300 mg loading dose Day 2-7: 75 mg orally once daily
  E.coli Endotoxin Day 7 - 2 ng/kg
  Interventions: Biological: Endotoxin; Drug: Clopidogrel
- No antiplatelet medication & Endotoxin (Placebo Comparator): No antiplatelet medication
  E.coli Endotoxin Day 7 - 2 ng/kg
  Interventions: Biological: Endotoxin
- Ticagrelor & Endotoxin (Experimental): Ticagrelor over 8 days (tablet) Day 1: 180 mg loading dose Day 2-7: 90 mg orally twice daily
  E.coli Endotoxin Day 7 - 2 ng/kg
  Interventions: Biological: Endotoxin; Drug: Ticagrelor

INTERVENTIONS:
Biological: Endotoxin — E.coli Endotoxin Day 7 - 2 ng/kg
  Other Names: E.coli Endotoxin
Drug: Clopidogrel — Clopidogrel (tablet) over 8 days Day 1: 300 mg loading dose Day 2-7: 75 mg orally once daily
  Arms: Clopidogrel & Endotoxin
Drug: Ticagrelor — Ticagrelor over 8 days (tablet) Day 1: 180 mg loading dose Day 2-7: 90 mg orally twice daily
  Other Names: Brilique
  Arms: Ticagrelor & Endotoxin

SUMMARY:
Platelets are the main type of blood cell involved in the formation of blood clots that cause heart attacks. The investigators give antiplatelet drugs (aspirin, for example) to reduce the risk of another clot forming in the future and causing another heart attack. Platelets are known to have a role in inflammation and infection as well as clotting. In a recent large clinical trial, known as the PLATO study, it was also shown that patients treated with a new antiplatelet medication (ticagrelor) developed fewer lung infections, as well as fewer heart attacks, compared to the current standard treatment (clopidogrel). The investigators would therefore like to investigate the reasons behind this and look at the effect of these medications on immune response. This may help us develop new drugs that have a better effect on immune response. The investigators are planning a clinical trial that investigates the effect of these medications on the immune response of healthy volunteers aged 18 to 65.

Only volunteers with no significant past medical history and not taking any medications will be included.

Thirty volunteers will receive either a normal dose of ticagrelor or clopidogrel or no antiplatelet medication for 1 week.

They will then attend the Sheffield Clinical Research Facility where their immune response will be stimulated using a safe, well established method. The investigators will do this with an injection of a low dose of endotoxin, which is part of the surface coating of some bacteria and has been used extensively in similar studies, in over a thousand volunteers over the past 20 years to investigate immune response. It is known to cause temporary flu-like symptoms that last approximately 68 hours. The investigators will take measurements of inflammatory markers, white blood cell function and platelet function and compare the effect of ticagrelor and clopidogrel on this immune response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, or female subjects not of childbearing potential (either surgically sterile or post menopausal)
* Age between 18 and 65 years inclusive
* Non smokers
* Body mass index (BMI) between 18 and 28 kg/m2 inclusive, with a body weight between 60-100 kg
* Subjects are to be in good health as determined by a medical history, physical examination, vital signs and clinical laboratory test results including renal and liver function and full blood count
* Subjects have given their informed consent before any trial-related activity

Exclusion Criteria:

* In the opinion of the investigator, subjects with, or a history of, cancer, diabetes or clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, haematological, dermatological, neurological, psychiatric, or other major disorders
* Subjects with a history of significant multiple drug allergies or with a known allergy to the study drugs or a medicine chemically related to the trial product
* Subjects who have had a clinically significant illness within 4 weeks of dosing
* Subjects taking regular medicines including NSAIDs, antibiotics, aspirin or anticoagulant therapy
* Any clinically significant abnormal laboratory test results at screening
* Subjects who have a supine blood pressure at screening, after resting for 5 minutes, higher than 150/90 mmHg or lower than 105/65 mmHg
* Subjects who have a supine heart rate at screening, after resting for 5 minutes, outside the range of 50-100 beats/min
* Subjects who have received any prescribed systemic or topical medication within two weeks prior to the start of dosing. Limited use of paracetamol or non-steroidal anti-inflammatory drugs (NSAIDs) prior to the initiation of the study will not necessarily require exclusion unless there is an ongoing requirement for these medications.
* Subjects who have received an investigational medicinal product within the previous four months (new chemical entity) or three months (licensed product) or subjects who have received a vaccine within three months preceding the start of dosing
* Subjects who have donated any blood or plasma in the month preceding the start of dosing
* Subjects who have a history of alcohol or drug abuse
* Subjects with mental incapacity or language barriers which preclude adequate understanding
* Subjects with a contraindication to ticagrelor (as listed in the SmPC - hypersensitivity to the active substance or any of its excipients, active pathological bleeding, history of intracranial hemorrhage, moderate to severe hepatic impairment and co-administration with strong CYP3A4 inhibitors)
* Subjects with a contraindication to clopidogrel (as listed in the SmPC - hypersensitivity to the active substance or any of its excipients, severe hepatic impairment, active pathological bleeding such as peptic ulcer or intracranial haemorrhage)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve of graph of C-reactive protein over time over 24 hours following administration of endotoxin | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robert Storey, Prof, Principal Investigator — University of Sheffield / Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Clinical Research Facility, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Derived] Thomas MR, Outteridge SN, Ajjan RA, Phoenix F, Sangha GK, Faulkner RE, Ecob R, Judge HM, Khan H, West LE, Dockrell DH, Sabroe I, Storey RF. Platelet P2Y12 Inhibitors Reduce Systemic Inflammation and Its Prothrombotic Effects in an Experimental Human Model. Arterioscler Thromb Vasc Biol. 2015 Dec;35(12):2562-70. doi: 10.1161/ATVBAHA.115.306528. Epub 2015 Oct 29. PMID 26515417